CLINICAL TRIAL: NCT00315094
Title: Prevention of Home Parenteral Nutrition (HPN) Infection, Depression and Improving Caregiving Problem Solving
Brief Title: Technological Home Care: Improving HPN Care With Videophone And Internet Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Carol Smith, RN, PhD, FAAN, Professor, School of Nursing, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 9655
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Home Parenteral Nutrition
Keywords: home parenteral nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Caregiving support interventions (FamTechCare)
- 2 (No Intervention): After a control period, this group crosses over to experimental interventions (Arm 1)

INTERVENTIONS:
Behavioral: Caregiving support interventions (FamTechCare) — One set of combined interventions to be tested in this study are nursing interventions for the prevention of catheter-related infection, reactive depression, and HPN home care problem-solving. The other set of combined interventions are for increasing social support and use of a short nap to reduce daily fatigue. Information about all the interventions were incorporated into Internet formats as a booster for reinforcement.
  Arms: 1

SUMMARY:
The purpose of this study is to help people with home parenteral nutrition (HPN) to avoid infections and feelings of depression or fatigue and to test how their health and quality of life change over time. Another purpose is to test the nurse teaching sessions and the method of obtaining support from the peer partner through videophone.

DETAILED DESCRIPTION:
Aim #1 Hypothesis

1. Dyad (patient-caregiver) participation in health care management and problem-solving method use with professionals will be greater in the experimental group than the control group
2. Dyad reactive depression will be lower in the experimental group than the control group
3. Dyad quality of life will be higher in the experimental group than the control group
4. Dyad health status scores will be higher and the dyad sleepiness scale will be lower in experimental group than the control group
5. Dyad Health Services Use will be lower in the experimental group than the control group
6. Catheter-related infections will be lower in the experimental than control patients

Aim #2 Hypotheses:

1. What is the cost of using the FamTechCare system compared to traditional care?
2. Is there a difference between efficiency scores of the experimental and control groups intervention, boosters and relative to dyads long-term health services use at 24 months?
3. What are the relationships among patient outcome variables and caregivers' rating of virtual nurse caring and caregiver adaption?
4. What are the relationships among use of FamTechCare, dyad participation in health care management scale score and dyad access to the Internet Weighted Score?

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Caregivers of HPN patients short- or long-term HPN
* able to participate in writing and other intervention activities
* able to speak/read/write English or Spanish

Exclusion Criteria:

* Patients with psychiatric disorders (e.g., schizophrenia, hallucinations) and physical disabilities that prevent use of intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Catheter related infection, depression, problem-solving and quality of life scores. | Experimental arm at T6, Control arm at T9.

SECONDARY OUTCOMES:
Ratings of virtual nurse caring | Experimental arm at T6, Control arm at T9.

CONTACTS AND LOCATIONS:
Overall Officials: Carol E Smith, PhD, RN, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States